CLINICAL TRIAL: NCT00240474
Title: A Comparison of Telmisartan 80 mg + Hydrochlorothiazide 12.5 mg With Amlodipine 10 mg + Hydrochlorothiazide 12.5 mg in the Control of Blood Pressure in Older Patients With Predominantly Systolic Hypertension. A Prospective, Randomised, Open-label, Blinded End-point Evaluation. (ATHOS Study)
Brief Title: A Comparison of Telmisartan + Hydrochlorothiazide With Amlodipine + Hydrochlorothiazide in the Control of Blood Pressure in Older Patients With Predominantly Systolic Hypertension (ATHOS Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.400
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; Amlodipine

INTERVENTIONS:
Drug: Telmisartan 80 mg + hydrochlorothiazide 12.5 mg
Drug: Amlodipine 10 mg + hydrochlorothiazide 12.5 mg

SUMMARY:
The primary objective of this study was test non-inferiority of telmisartan 80 mg + hydrochlorothiazide (HCTZ) 12.5 mg in comparison to amlodipine 10 mg + HCTZ 12.5 mg in reducing ambulatory systolic blood pressure (SBP) in the last 6 hours of the 24-hour dosing interval (determined by ambulatory blood pressure monitoring: ABPM) in elderly patients with predominantly systolic hypertension.

ELIGIBILITY:
Inclusion criteria:

* aged at least 60 years old
* mean SBP greater than 140 mmHg and mean DBP less than or equal to 95 mmHg
* 24-hour mean ambulatory SBP greater than 125 mmHg
* hypertensive patients not on current antihypertensive therapy or able to stop their current treatment for a period of up to eighteen weeks
* willing and able to provide written informed consent

Exclusion criteria:

* women of child-bearing potential who are NOT practicing acceptable means of birth control
* known or suspected secondary hypertension
* mean SBP equal to or greater than 200 mmHg
* hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  * bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, patients post-renal transplant or with only one functioning kidney
  * clinically relevant hypokalemia or hyperkalemia
  * uncorrected volume or sodium depletion
* primary aldosteronism
* hereditary fructose intolerance
* biliary obstructive disorders
* patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin-II receptor antagonists
* history of drug or alcohol dependency within the previous six months
* chronic administration of any medication known to affect blood pressure, other than the trial medication
* concurrent participation in another clinical trial or any investigational therapy within thirty days prior to signing the consent form.
* symptomatic congestive heart failure (New York Heart Academy (NYHA) functional class CHF II-IV)
* unstable angina pectoris, myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) surgery less than three months prior to informed consent
* stroke less than six months prior to informed consent
* sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant arrhythmias as determined by the investigator
* hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve
* insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for the previous three months
* night-shift workers who routinely sleep during the daytime and whose working hours include midnight to 4:00 AM
* known allergic hypersensitivity to any component of the formulations under investigation
* concomitant therapy with lithium, cholestyramine or colestipol resins. non-compliance with study medication (defined as less than 80% or more than 120%) during the run-in period
* current treatment with any antihypertensive agent
* any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan, amlodipine or hydrochlorothiazide

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-12; Primary Completion 2004-03 (Actual); Study Completion 2004-03

PRIMARY OUTCOMES:
Change from baseline in the last 6-hour mean (relative to dose time) in SBP as measured by 24-hour ABPM at the end-of-study visit | 14 weeks

SECONDARY OUTCOMES:
Change from baseline in DBP in the last six hours of the 24-hour dose period | week 8 and 14
Change from baseline in pulse pressure (PP) in the last six hours of the 24-hour dose period | week 8 and 14
Change from baseline SBP and DBP for other time intervals ( i.e. 24-hour mean, morning mean (06:00-11:59), daytime mean (06:00-21:59), and night-time mean (22:00-05:59)) | week 8 and 14
Change from baseline in patient HRQL as measured by the Psychological General Well-Being (PGWB) index. | week 8 and 14
Change from baseline in SBP in the last six hours of the 24-hour dose period (as measured by 24-hour ABPM). | 8 weeks
Proportion of patients achieving a target response in SBP | 14 weeks
Proportion of patients achieving SBP control | 14 weeks
Proportion of patients achieving normal blood pressure | 14 weeks
Proportion of patients achieving high-normal blood pressure | 14 weeks
Change from baseline in trough seated SBP | 14 weeks
Change from baseline in trough seated DBP | 14 weeks
Safety and tolerability of the combination of telmisartan 80 mg and HCTZ 12.5 mg compared with amlodipine 10 mg and HCTZ 12.5 mg | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BIL UK / Ireland
Locations (72):
- Belgium (4):
  - A.C.Z. Antwerpen/Stuyvenberg, Antwerp
  - Boehringer Ingelheim Investigational Site, Aywaille
  - A.Z. VUB, Brussels
  - C.H.U. Liège (Ourthe-Amblève), Esneux
- Denmark (10):
  - Boehringer Ingelheim Investigational Site, Aabenraa
  - Boehringer Ingelheim Investigational Site, Christiansfeld
  - Boehringer Ingelheim Investigational Site, Haderslev
  - Boehringer Ingelheim Investigational Site, Herning
  - Boehringer Ingelheim Investigational Site, Hvidovre
  - Boehringer Ingelheim Investigational Site, Odder
  - Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - Boehringer Ingelheim Investigational Site, Vildberg
  - Boehringer Ingelheim Investigational Site, Vildbjerg
  - Boehringer Ingelheim Investigational Site, Vinderup
- Finland (6):
  - Hämeenlinnan lääkäriasema Oy, Linnan klinikka, Hämeenlinna
  - Diacor, Helsinki
  - Kiljava Medical Research, Hyvinkää
  - Boehringer Ingelheim Investigational Site, Jyväskylä
  - Kouvolan lääkäriasema, Kouvola
  - Hatanpään terveyskeskussairaala, Tampere
- France (6):
  - Boehringer Ingelheim Investigational Site, Angers
  - Boehringer Ingelheim Investigational Site, Aÿ
  - Boehringer Ingelheim Investigational Site, Château Gontier Bazougues
  - Boehringer Ingelheim Investigational Site, Jarny
  - Hôpital de la Timone, Marseille
  - Boehringer Ingelheim Investigational Site, Mayenne
- Germany (21):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Ellefeld
  - Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Flörsheim
  - Boehringer Ingelheim Investigational Site, Hagen
  - Boehringer Ingelheim Investigational Site, Hatten
  - Boehringer Ingelheim Investigational Site, Kelkheim
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site, Marl
  - Boehringer Ingelheim Investigational Site, Münster
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Ornbau
  - Boehringer Ingelheim Investigational Site, Rednitzhembach
  - Boehringer Ingelheim Investigational Site, Riesa
  - Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - Boehringer Ingelheim Investigational Site, Straßkirchen
  - Boehringer Ingelheim Investigational Site, Wallerfing
  - Boehringer Ingelheim Investigational Site, Werne
  - Boehringer Ingelheim Investigational Site, Westerkappeln
  - Deutsche Klinik für Diagnostik GmbH, Wiesbaden
  - Evangelisches Krankenhaus, Witten
- Ireland (6):
  - 19 Redwood View, Dublin
  - Adelaide and Meath Hospitals (incorrporating NCH), Dublin
  - Boehringer Ingelheim Investigational Site, Dublin
  - Cardioperfect Research Room, Dublin
  - Beaumont Park Clinic, Dublin
  - Boehringer Ingelheim Investigational Site, Kilkenny
- Italy (6):
  - Ospedale S. Luigi - S. Currò, Catania
  - Università di Ferrara, Ferrara
  - Az. Osped. Universitaria "Osp. Riuniti", Foggia
  - Azienda Ospedaliera "Maggiore della Carità", Novara
  - Ospedale Scillesi d'America, Scilla (rc)
  - Ospedale Civile, Vittorio Veneto (TV)
- Netherlands (9):
  - Boehringer Ingelheim Investigational Site, Beek en Donk
  - Boehringer Ingelheim Investigational Site, Ewijk
  - Boehringer Ingelheim Investigational Site, Musselkanaal
  - Boehringer Ingelheim Investigational Site, Oude Pekela
  - Boehringer Ingelheim Investigational Site, Rijswijk
  - Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - Boehringer Ingelheim Investigational Site, The Hague
  - Boehringer Ingelheim Investigational Site, Vaals
  - Boehringer Ingelheim Investigational Site, Voerendaal
- Boehringer Ingelheim Investigational Site, Pretoria, South Africa
- Spain (3):
  - Avda. Menendez Pidal, s&n, Córdoba
  - Hospital Gral de Jerez de la Frontera, Jerez de La Frontera / Cádiz
  - Cardiology Service, Santander